CLINICAL TRIAL: NCT02977650
Title: EUS-FNA for Patients Taking Anticoagulants Without Heparin Bridge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hokkaido Pancreatobiliary Endoscopic Intervention Study Group (Network)
Responsible Party: Principal Investigator, Kazumichi Kawakubo, M.D., Ph.D., Hokkaido Pancreatobiliary Endoscopic Intervention Study Group
Other Study IDs: 016-0040
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Endoscopic Ultrasonography-guided Fine Needle Aspiration
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic ultrasonography-guided fine needle aspiration
  Other Names: EUS-FNA

SUMMARY:
To evaluate the feasibility of EUS-FNA for patients taking anticoagulants without heparin bridge.

ELIGIBILITY:
Inclusion Criteria:

* Taking anticoagulants
* Written informed consent

Exclusion Criteria:

* Platelets count less than 50000/μl
* PT-INR more than 2.6
* ASA more than 3
* Severe bleeding tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking anticoagulants who underwent EUS-FNA
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The rate of bleeding adverse events | Within 2 weeks

SECONDARY OUTCOMES:
The rate of thromboembolic events | Within 2 weeks
The rate of other adverse events | Within 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Undecided